CLINICAL TRIAL: NCT05385276
Title: Transverse Supraumbilical Versus Pfannenstiel Incision For Cesarean Section In Morbidly Obese Women "A Randomized Controlled Trial"
Brief Title: Transverse Supraumbilical Versus Pfannenstiel Incision For Cesarean Section In Morbidly Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Arafa, Principal Investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07052022
Record Dates: First submitted 2022-05-07; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse supraumbilical incision (Experimental): The skin incision will be performed as a straight transverse skin incision 3-5cm above the umbilicus after maximum retraction of the panniculus caudally using two towel clips, to facilitate the approach to the lower uterine segment.
  Interventions: Procedure: Transverse supraumbilical incision
- Pfannenstiel Incision (Experimental): The skin incision is a transverse upward concavity, typically initiated two finger breadths above the symphysis pubis and extended in the direction of the anterior superior iliac spine below and medial to it about (2 - 3 cm).
  Interventions: Procedure: Pfannenstiel Incision

INTERVENTIONS:
Procedure: Transverse supraumbilical incision — The skin incision will be performed as a straight transverse skin incision 3-5cm above umbilicus after maximum retraction the panniculus caudally using two towel clips, to facilitate the approach to the lower uterine segment The skin incision is a transverse upward concavity, typically initiated two finger-breadths above the symphysis pubis and extended in the direction of the anterior superior iliac spine below and medial to it about (2 - 3 cm) .
  Arms: Transverse supraumbilical incision
Procedure: Pfannenstiel Incision — The skin incision is a transverse upward concavity, typically initiated two finger-breadths above the symphysis pubis and extended in the direction of the anterior superior iliac spine below and medial to it about (2 - 3 cm).
  Arms: Pfannenstiel Incision

SUMMARY:
cesarean section is one of the most common operative procedures performed in modern obstetrics, that become increasingly common in both developed and developing countries for a variety of reasons today, thus any useful refinement in the operative technique, however minimal, is likely to yield substantial benefits.

In morbidly obese women with a panniculus, the supraumbilical incision is a new technique that showed definite advantages over the Pfannenstiel incision that will avoid burying the wound under a large panniculus and affords excellent abdominal exposure, less blood loss, less post-operative pain, earlier ambulation, and shorter hospital stay. All these advantages were attributed to minimal tissue manipulation.

DETAILED DESCRIPTION:
The prevalence of obesity has reached pandemic proportions across nations. Morbid obesity has a dramatic impact on pregnancy outcomes. Cesarean section in these women poses many surgical, anesthetic, and logistical challenges.

The rapid upswing in obesity prevalence across nations, ages, and ethnic groups has reached alarming and pandemic proportions.

The prevalence of morbid obesity (BMI>40 kg/m2) has increased by 50% between 2000 and 2005, with 8% of women in the reproductive age group being morbidly obese.

The percentage of women with a body mass index (BMI) of 50 Kg/m2 or more has increased five-fold in 20 years. Obesity is currently the most prevalent health threat the world over and its influence on general health is rapidly increasing.

The incidence of pregnancy-related pathology is higher in obese patients. Obstetricians are often confronted with difficult decisions when such patients are about to give birth. Indeed, in obese patients, labor is induced twice as frequently and vaginal delivery has to be interrupted more frequently due to an abnormal fetal heart rate or fetopelvic disproportion.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with morbid obesity (BMI > 40)
* Patients with an abdominal panniculus covering the supra pubic skin crease.
* Patients with a singleton pregnancy.
* All indications for elective cesarean section.
* Hemoglobin ≥ 10 g/dl.
* Since obesity is a disease associated commonly with co-morbidities such as diabetes mellitus, hypertension and sometimes chest problem these conditions will not be excluded, despite being significant factors that may affect wound healing and this will be analyzed in subgroups.
* Preoperative glycemic control (HbA1C level < 7 percent) for women with diabetes.

Exclusion Criteria:

* Antepartum Hemorrhage and placenta previa (more bleeding and operative time anticipated will interfere with the interpretation of operative date)
* Drugs intake that affects bleeding or tissue healing e.g., anti-coagulants, immunosuppressive drugs and chronic use of steroids (more than 14 days pre-operative).
* Multiple gestation (higher blood loss is anticipated).
* Patients diagnosed with intra amniotic infections (infections increases bleeding and incidence for post-operative infections).
* Patients with (HELLP syndrome) hemolysis, elevated liver enzymes and low platelets or bleeding disorders (the need for blood and blood products is higher than average).
* Patients with bleeding disorders or auto immune diseases (both affects bleeding and time needed for hemostasis as well as tissue healing).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean operative time | during the procedure
  measurement of intra-operative times in minutes

SECONDARY OUTCOMES:
Mean Intra-operative blood loss | during the procedure
  By comparing pre-operative Hemoglobin with values taken 24 hours after the operation.
Occurrence of Post-operative Surgical site infection | 7 days
  The participants will be scheduled for a return visit after 7 days for removal of the sutures and recording of any signs of surgical site infection (hotness, tenderness, exudation, pus discharge).
Occurrence of surgical complications | during the operation
  observation of intraoperative visceral or vascular injuries
Mean hospital stay | 3 days postoperatively
  The time between the operation and discharge from hospital
VAS score of pain | 24 hours
  The severity of postoperative pain was assessed using the Visual Analogue Scale (VAS will be evaluated postoperatively and every 2 hours during the first 6 hours and then every 6 hours for the next 24 hours postoperatively).
  VAS is a 0 -10 scale in which 0 means that the patient feels no pain and 10 means that the patient is in maximal pain.
Mean Intra-operative blood loss | During the procedure
  comparing pre-operative Hematocrit values with values taken 24 hours after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamed, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No